CLINICAL TRIAL: NCT07195643
Title: Predictive Factors of Drain Insertion After Laparoscopic Cholecystectomy: A Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mohammedsadeq A. Shweliya, Principal Investigator, College of Medicine, University of Baghdad, University of Baghdad
Other Study IDs: Drainage after cholecystectomy
Record Dates: First submitted 2025-08-20; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cholecystitis
Keywords: Laproscopic cholecystectomy; Drain; Predictive factors
MeSH Terms: conditions — Cholecystitis | interventions — Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent laparoscopic cholecystectomy: This study cohort consists of 559 patients who underwent laparoscopic cholecystectomy (LC) at Safeer Al-Husain Hospital, Karbala, Iraq, between January 2025 and March 2025. Patients were included regardless of age, gender, body mass index, or gallbladder pathology, as long as they underwent elective or emergency LC.
  Interventions: Other: Drain

INTERVENTIONS:
Other: Drain — We want to put a assess the predictive factors for prophylactic drain after cholecystectomy.

SUMMARY:
This study looks at when surgical drains are truly needed after laparoscopic gallbladder removal (laparoscopic cholecystectomy). Drains are sometimes placed during surgery to prevent fluid buildup or infection, but many studies show they are not always necessary. We reviewed 559 patients who had this surgery at Safeer Al-Husain Hospital in Karbala, Iraq. The goal of this study is to help doctors decide more carefully when to use drains, so patients can avoid unnecessary tubes and recover more quickly.

DETAILED DESCRIPTION:
Background:

Laparoscopic cholecystectomy (LC) is the standard treatment for symptomatic gallstones, offering benefits such as reduced pain, shorter hospital stays, and faster recovery. However, postoperative complications like bile leakage, hemorrhage, and infection remain concerns. Many surgeons use intraoperative drains routinely to prevent these complications, though evidence increasingly suggests selective use may be preferable. Few studies have systematically identified which patient or intraoperative factors predict the need for drain placement.

Objective:

To identify demographic, clinical, and intraoperative predictors of surgical drain placement after LC, enabling evidence-based, selective drain use.

Methods:

* Design: prospective cross-sectional study at Safeer Al-Husain Hospital, Karbala, Iraq.
* Population: 559 patients undergoing LC.
* Data Collection: Patient demographics, operative details, intraoperative findings, and drain usage were extracted from standardized hospital records.
* Statistical Analysis: Associations between patient/surgical variables and drain placement were assessed using univariate and multivariate logistic regression. Statistical significance was defined as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Underwent laparoscopic cholecystectomy (LC) at Safeer Al-Husain Hospital, Karbala, Iraq.
* Both male and female patients.
* Diagnosed with gallstone disease, including:

  * Chronic cholecystitis
  * Acute cholecystitis
  * Acute-on-chronic cholecystitis
  * Biliary colic

Exclusion Criteria:

* Conversion from laparoscopic to open cholecystectomy prior to completion of the procedure.
* Patients undergoing emergency surgery for gallbladder perforation with generalized peritonitis, where standard laparoscopic cholecystectomy was not feasible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients who underwent laparoscopic cholecystectomy at Safeer Al-Husain Hospital, Karbala, Iraq. Both male and female patients with gallstone disease (chronic cholecystitis, acute cholecystitis, acute-on-chronic cholecystitis, or biliary colic) were included. This cohort represents a typical Middle Eastern surgical population treated in a tertiary referral hospital, with a wide range of demographic and clinical characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients undergoing laparoscopic cholecystectomy who require intraoperative drain insertion | Immediately post-op, day zero

SECONDARY OUTCOMES:
Operative time | Day 0 (intraoperative period)
  Duration of laparoscopic cholecystectomy measured in minutes, from first incision to closure
Incidence of intraoperative bile or stone spillage | Day 0 (intraoperative period)
  Documented occurrence of bile leakage or gallstone spillage during the procedure.
Gallbladder wall thickness | Baseline (preoperative imaging)
  Preoperative ultrasound measurement of gallbladder wall thickness and its association with drain placement.
Presence of adhesions | Day 0 (intraoperative period)
  Intraoperative finding of pericholecystic or omental adhesions
Patient demographics | Baseline (before surgery)
  Age, Gender (male/female), Body Mass Index,
Clinical presentation | Baseline (preoperative assessment)
  Acute inflammation, chronic inflammation, biliary colic, acute on chronic inflammation
Trocar insertion technique | Intraoperative
  Easy blind, difficult blind, easy open, difficult open, or Veress needle.
Gallbladder anatomy | Intraoperative
  Classical, adhesions, anomaly
Common bile duct anatomy | Intraoperative
Number of clips used | Intraoperative
Hepatic bed status | Intraoperative
  None, oozing, active bleeding
Gallbladder extraction technique | Intraoperative
  Without manipulation, evacuation of content, wound extension, extension + evacuation, endobag
Other adverse events | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Arkan Shubber AbdulKhaliq Al-hamdany, F.I.B.M.S., Study Director — Iraqi Ministry of Health, Karbala Health Directorate
Locations (1):
- Safeer Al-Husain Hospital, Karbala, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu H, Liu D, Zhou D, Wu J, Yu Y, Jin Y, Ye D, Ding C, Zhang X, Huang B, Peng S, Li J. Effectiveness of no drainage after elective day-case laparoscopic cholecystectomy, even with intraoperative gallbladder perforation: a randomized controlled trial. Langenbecks Arch Surg. 2023 Mar 1;408(1):112. doi: 10.1007/s00423-023-02846-z. PMID 36856748
- [Background] Xu M, Tao YL. Drainage versus No Drainage after Laparoscopic Cholecystectomy for Acute Cholecystitis: A Meta-Analysis. Am Surg. 2019 Jan 1;85(1):86-91. PMID 30760351
- [Background] Bawahab MA, Abd El Maksoud WM, Alsareii SA, Al Amri FS, Ali HF, Nimeri AR, Al Amri AR, Assiri AA, Abdul Aziz MI. Drainage vs. non-drainage after cholecystectomy for acute cholecystitis: a retrospective study. J Biomed Res. 2014 May;28(3):240-5. doi: 10.7555/JBR.28.20130095. Epub 2014 Apr 10. PMID 25013408
- [Background] Calini G, Brollo PP, Quattrin R, Bresadola V. Predictive Factors for Drain Placement After Laparoscopic Cholecystectomy. Front Surg. 2022 Feb 2;8:786158. doi: 10.3389/fsurg.2021.786158. eCollection 2021. PMID 35187046